CLINICAL TRIAL: NCT02981368
Title: A PrOspective Phase 2/3 Multi-Center Study of 18F-DCFPyL PET/CT Imaging in Patients With PRostate Cancer: Examination of Diagnostic AccuracY (OSPREY)
Brief Title: Study of 18F-DCFPyL PET/CT Imaging in Patients With Prostate Cancer
Acronym: OSPREY
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PyL 2301
Record Dates: First submitted 2016-11-22; First posted 2016-12-05 (Estimated); Results first posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Prostate Cancer
Keywords: Diagnostic; Imaging; 2301; PET/CT; PyL; PSMA; radical prostatectomy; metastatic prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Disease | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18F-DCFPyL Injection (Experimental): 9±1 mCi (333±37 MBq) IV injection of 18F-DCFPyL
  Interventions: Drug: 18F-DCFPyL Injection; Diagnostic Test: PET/CT imaging

INTERVENTIONS:
Drug: 18F-DCFPyL Injection — A single dose of 9±1 mCi (333±37 MBq) IV injection of 18F-DCFPyL
  Other Names: PyL
Diagnostic Test: PET/CT imaging — PET/CT imaging will be acquired 1-2 hours post-PyL injection

SUMMARY:
This study evaluates the safety and diagnostic performance of 18F-DCFPyL Injection in patients with at least high risk prostate cancer who are planned for radical prostatectomy with lymphadenectomy (Cohort A) or in patients with locally recurrent or metastatic disease willing to undergo biopsy (Cohort B).

Cohort B is complete and no longer recruiting subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate.
2. Subjects provide signed informed consent and confirm that they are able and willing to comply with all protocol requirements.

Cohort A Only:

* At least high risk prostate cancer defined by NCCN Guidelines Version 3.2016 (clinical stage ≥T3a or PSA >20 ng/mL or Gleason score ≥8).
* Scheduled or planned radical prostatectomy with PLND.

Cohort B Only: [Enrollment is complete; No longer recruiting subjects]

* Radiologic evidence of local recurrence or new or progressive metastatic disease demonstrated on anatomical imaging (CT, MRI, or ultrasound), whole-body bone scan (99m-Tc-MDP or Na-18F) within 4 weeks of enrollment.
* If prior treatment with radiation or ablative therapy, evidence of recurrence outside the confines of prior treated site(s) is needed.
* Scheduled or planned percutaneous biopsy of at least one amenable lesion.

Exclusion Criteria:

1. Subjects administered any high energy (>300 KeV) gamma-emitting radioisotope within five physical half-lives, or any IV iodinated contrast medium within 24 hours, or any high density oral contrast medium (oral water contrast is acceptable) within 5 days, prior to study drug injection.
2. Subjects with any medical condition or other circumstance that, in the opinion of the investigator, compromise obtaining reliable data, achieving study objectives, or completion.

Cohort A Only:

* Patients with prior androgen deprivation therapy or any investigational neoadjuvant agent or intervention

Cohort B Only: [Enrollment is Complete; No longer recruiting subjects]

* Prior radiation or ablative therapy to intended site of biopsy, if within the prostate bed
* Initiation of new therapy for recurrent and/or progressive metastatic disease since radiographic documentation of recurrence/progression.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Morris, MD, Study Chair — Memorial Sloan Kettering Cancer Center; Kenneth J Pienta, MD, Principal Investigator — Johns Hopkins University
Locations (10):
- United States (8):
  - University of California at San Francisco (UCSF) - Mt. Zion Hospital, San Francisco, California
  - Yale University Department of Radiology and Biomedical Imaging, New Haven, Connecticut
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Washington University Mallinckrodt Institute of Radilogy, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
- Canada (2):
  - Jewish General Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec (CHUQ), Québec

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- High Risk Prostate Cancer (Cohort A): Patients with high risk prostate cancer planned for radical prostatectomy with pelvic lymph node dissection were enrolled to receive a single dose of 9 mCi (333 MBq) IV injection of 18F-DCFPyL, followed by PET/CT imaging acquired 1-2 hours post-PyL injection.
- Recurrent or Metastatic Prostate Cancer (Cohort B): Patients with presumptive radiologic evidence of prostate cancer recurrence or metastasis on conventional imaging and planned for conventional image-guided biopsy were enrolled to receive a single dose of 9 mCi (333 MBq) IV injection of 18F-DCFPyL, followed by PET/CT imaging acquired 1-2 hours post-PyL injection.
Period: Overall Study
Arm/Group | High Risk Prostate Cancer (Cohort A) | Recurrent or Metastatic Prostate Cancer (Cohort B)
Started | 268 | 117
Completed | 248 | 102
Not Completed | 20 | 15

BASELINE CHARACTERISTICS:
Population: Safety population; total number of patients who received 18F-DCFPyL injection.
Groups:
- Total: Total of all reporting groups
Arm/Group | High Risk Prostate Cancer (Cohort A) | Recurrent or Metastatic Prostate Cancer (Cohort B) | Total
Number analyzed (Participants) | 268 | 117 | 385
Age, Continuous [Median (Full Range); unit: years] | 65 [46 to 84] | 68 [45 to 86] | 66 [45 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 268 | 117 | 385
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 233 | 101 | 334
  Race: Black or African American | 23 | 6 | 29
  Race: Asian | 7 | 4 | 11
  Race: Other | 2 | 3 | 5
  Race: Unknown or Not Reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Specificity of 18F-DCFPyL PET/CT Imaging to Detect Metastatic Prostate Cancer Within the Pelvic Lymph Nodes Relative to Histopathology in High Risk Prostate Cancer Participants (Cohort A)
Description: The primary analysis in Cohort A will test the co-primary endpoints of sensitivity and specificity of 18F-DCFPyL PET/CT imaging relative to histopathology for metastatic disease in pre-prostatectomy patients. For each co-primary endpoint there will be three independent imaging readers. At least two of the three readers must reject the null hypothesis for specificity to be deemed a success. If specificity is a success, then the same two readers need to reject the null hypothesis for sensitivity to reach overall success of the primary endpoint.
Time Frame: Within 28 days of imaging, radical prostatectomy with pelvic lymph node dissection will occur.
Population: The Evaluable Set of high risk prostate cancer participants (Cohort A) includes those who received 18F-DCFPyL, had a prostatectomy or lymphadenectomy, and provided a 18F-DCFPyL PET/CT image result and a corresponding histopathology result.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- High Risk Prostate Cancer (Cohort A): High risk prostate cancer participants planned for radical prostatectomy with pelvic lymph node dissection were enrolled to receive a single dose of 9 mCi (333 MBq) IV injection of 18F-DCFPyL, followed by PET/CT imaging acquired 1-2 hours post-PyL injection.
Arm/Group | High Risk Prostate Cancer (Cohort A)
Number analyzed (Participants) | 252
percentage of participants
  Central Reader 1 | 97.9 [94.52 to 99.37]
  Central Reader 2 | 98.9 [96.00 to 99.96]
  Central Reader 3 | 96.3 [93.64 to 98.99]

2. Primary Outcome: Sensitivity of 18F-DCFPyL PET/CT Imaging to Detect Metastatic Prostate Cancer Within the Pelvic Lymph Nodes Relative to Histopathology in High Risk Prostate Cancer Participants (Cohort A)
Description: as for outcome 1
Time Frame: Within 28 days of imaging, radical prostatectomy with pelvic lymph node dissection will occur.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High Risk Prostate Cancer (Cohort A)
Number analyzed (Participants) | 252
percentage of participants
  Central Reader 1 | 41.9 [29.65 to 54.22]
  Central Reader 2 | 30.6 [19.17 to 42.12]
  Central Reader 3 | 40.3 [28.11 to 52.53]

3. Secondary Outcome: Shift From Baseline in Selected Hematology Laboratory Values at Follow-up (Safety Outcome Measure)
Description: Shifts from baseline to worst post-baseline visit for hematology laboratory values for all participants included in the Safety Set. The Safety Set includes all participants who received any amount of 18F-DCFPyL. Data are presented for participants in Cohort A and Cohort B.
Time Frame: From time of screening (baseline) until pre-surgery/biopsy (within 28 days post-study drug dosing).
Population: The Safety Set includes all participants who received any amount of 18F-DCFPyL.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A - Follow-up Value: Low: Cohort A participants who had a follow-up laboratory value that was below the lower limit of normal. Cohort A were high risk cancer participants planned for radical prostatectomy with pelvic lymph node dissection.
- Cohort B - Follow-up Value: Low: Cohort B participants who had a follow-up laboratory value that was below the lower limit of normal. Cohort B were participants with presumptive radiologic evidence of prostate cancer recurrence or metastasis on conventional imaging and planned for conventional image-guided biopsy.
- Cohort A - Follow-up Value: Normal: Cohort A participants who had a follow-up laboratory value that was within normal limit. Cohort A were high risk cancer participants planned for radical prostatectomy with pelvic lymph node dissection.
- Cohort B - Follow-up Value Normal: Cohort B participants who had a follow-up laboratory value that was within normal limits. Cohort B were participants with presumptive radiologic evidence of prostate cancer recurrence or metastasis on conventional imaging and planned for conventional image-guided biopsy.
- Cohort A - Follow-up Value: High: Cohort A participants who had a follow-up laboratory value that was above the upper limit of normal. Cohort A were high risk cancer participants planned for radical prostatectomy with pelvic lymph node dissection.
- Cohort B - Follow-up Value: High: Cohort B participants who had a follow-up laboratory value that was above the upper limit of normal. Cohort B were participants with presumptive radiologic evidence of prostate cancer recurrence or metastasis on conventional imaging and planned for conventional image-guided biopsy.
- Cohort A - Follow-up Value: Missing: Cohort A participants who did not have a follow-up laboratory value. Cohort A were high risk cancer participants planned for radical prostatectomy with pelvic lymph node dissection.
- Cohort B - Follow-up Value: Missing: Cohort B participants who did not have a follow-up laboratory value. Cohort B were participants with presumptive radiologic evidence of prostate cancer recurrence or metastasis on conventional imaging and planned for conventional image-guided biopsy.
Arm/Group | Cohort A - Follow-up Value: Low | Cohort B - Follow-up Value: Low | Cohort A - Follow-up Value: Normal | Cohort B - Follow-up Value Normal | Cohort A - Follow-up Value: High | Cohort B - Follow-up Value: High | Cohort A - Follow-up Value: Missing | Cohort B - Follow-up Value: Missing
Number analyzed (Participants) | 268 | 117 | 268 | 117 | 268 | 117 | 268 | 117
Participants
  Hematocrit: number analyzed (Participants) | 55 | 32 | 197 | 53 | 2 | 0 | 14 | 32
  Hematocrit: Cohort A - Baseline Value: Low | 26 | 0 | 12 | 0 | 0 | 0 | 2 | 0
  Hematocrit: Cohort B - Baseline Value: Low | 0 | 31 | 0 | 6 | 0 | 0 | 0 | 10
  Hematocrit: Cohort A - Baseline Value: Normal | 29 | 0 | 179 | 0 | 1 | 0 | 12 | 0
  Hematocrit: Cohort B - Baseline Value: Normal | 0 | 1 | 0 | 47 | 0 | 0 | 0 | 22
  Hematocrit: Cohort A - Baseline Value: High | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0
  Hematocrit: Cohort B - Baseline Value: High | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit: Cohort A - Baseline Value: Missing | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Hematocrit: Cohort B - Baseline Value: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin: number analyzed (Participants) | 34 | 35 | 218 | 50 | 2 | 0 | 14 | 32
  Hemoglobin: Cohort A - Baseline Value: Low | 16 | 0 | 3 | 0 | 0 | 0 | 2 | 0
  Hemoglobin: Cohort B - Baseline Value: Low | 0 | 33 | 0 | 6 | 0 | 0 | 0 | 13
  Hemoglobin: Cohort A - Baseline Value: Normal | 18 | 0 | 210 | 0 | 1 | 0 | 11 | 0
  Hemoglobin: Cohort B - Baseline Value: Normal | 0 | 2 | 0 | 43 | 0 | 0 | 0 | 18
  Hemoglobin: Cohort A - Baseline Value: High | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 0
  Hemoglobin: Cohort B - Baseline Value: High | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Hemoglobin: Cohort A - Baseline Value: Missing | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Cohort B - Baseline Value: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: number analyzed (Participants) | 16 | 12 | 237 | 72 | 1 | 1 | 14 | 32
  Platelets: Cohort A - Baseline Value: Low | 12 | 0 | 3 | 0 | 0 | 0 | 1 | 0
  Platelets: Cohort B - Baseline Value: Low | 0 | 9 | 0 | 2 | 0 | 0 | 0 | 3
  Platelets: Cohort A - Baseline Value: Normal | 4 | 0 | 230 | 0 | 1 | 0 | 13 | 0
  Platelets: Cohort B - Baseline Value: Normal | 0 | 3 | 0 | 70 | 0 | 0 | 0 | 29
  Platelets: Cohort A - Baseline Value: High | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Platelets: Cohort B - Baseline Value: High | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Platelets: Cohort A - Baseline Value: Missing | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Platelets: Cohort B - Baseline Value: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocytes: number analyzed (Participants) | 49 | 42 | 205 | 42 | 0 | 1 | 14 | 32
  Erythrocytes: Cohort A - Baseline Value: Low | 29 | 0 | 8 | 0 | 0 | 0 | 2 | 0
  Erythrocytes: Cohort B - Baseline Value: Low | 0 | 36 | 0 | 1 | 0 | 0 | 0 | 10
  Erythrocytes: Cohort A - Baseline Value: Normal | 20 | 0 | 194 | 0 | 0 | 0 | 11 | 0
  Erythrocytes: Cohort B - Baseline Value: Normal | 0 | 6 | 0 | 39 | 0 | 0 | 0 | 22
  Erythrocytes: Cohort A - Baseline Value: High | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Erythrocytes: Cohort B - Baseline Value: High | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
  Erythrocytes: Cohort A - Baseline Value: Missing | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Erythrocytes: Cohort B - Baseline Value: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes: number analyzed (Participants) | 11 | 7 | 220 | 75 | 23 | 3 | 14 | 32
  Leukocytes: Cohort A - Baseline Value: Low | 7 | 0 | 3 | 0 | 0 | 0 | 2 | 0
  Leukocytes: Cohort B - Baseline Value: Low | 0 | 7 | 0 | 1 | 0 | 0 | 0 | 2
  Leukocytes: Cohort A - Baseline Value: Normal | 4 | 0 | 208 | 0 | 18 | 0 | 12 | 0
  Leukocytes: Cohort B - Baseline Value: Normal | 0 | 0 | 0 | 71 | 0 | 1 | 0 | 30
  Leukocytes: Cohort A - Baseline Value: High | 0 | 0 | 7 | 0 | 5 | 0 | 0 | 0
  Leukocytes: Cohort B - Baseline Value: High | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 0
  Leukocytes: Cohort A - Baseline Value: Missing | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Leukocytes: Cohort B - Baseline Value: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Shift From Baseline in Selected Clinical Chemistry Laboratory Values at Follow-up (Safety Outcome Measure)
Description: Shifts from baseline to worst post-baseline visit for clinical chemistry laboratory values for all participants included in the Safety Set. The Safety Set includes all participants who received any amount of 18F-DCFPyL. Data are presented for participants in Cohort A and Cohort B.
Time Frame: From time of screening (baseline) until pre-surgery/biopsy (within 28 days post-study drug dosing).
Population: The Safety Set includes all participants who received any amount of 18F-DCFPyL.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort B - Follow-up Value: Low: Cohort B participants who had a follow-up laboratory value that was below the lower limit of normal. Cohort B were participants with presumptive radiologic evidence of prostate cancer recurrence or metastasis on conventional imaging and planned conventional image-guided biopsy.
- Cohort B - Follow-up Value: Normal: Cohort B participants who had a follow-up laboratory value that was within normal limits. Cohort B were participants with presumptive radiologic evidence of prostate cancer recurrence or metastasis on conventional imaging and planned conventional image-guided biopsy.
- Cohort B - Follow-up Value: High: Cohort B participants who had a follow-up laboratory value that was above the upper limit of normal. Cohort B were participants with presumptive radiologic evidence of prostate cancer recurrence or metastasis on conventional imaging and planned conventional image-guided biopsy.
- Cohort B - Follow-up Value: Missing: Cohort B participants who did not have a follow-up laboratory value. Cohort B were participants with presumptive radiologic evidence of prostate cancer recurrence or metastasis on conventional imaging and planned conventional image-guided biopsy.
Arm/Group | Cohort A - Follow-up Value: Low | Cohort B - Follow-up Value: Low | Cohort A - Follow-up Value: Normal | Cohort B - Follow-up Value: Normal | Cohort A - Follow-up Value: High | Cohort B - Follow-up Value: High | Cohort A - Follow-up Value: Missing | Cohort B - Follow-up Value: Missing
Number analyzed (Participants) | 268 | 117 | 268 | 117 | 268 | 117 | 268 | 117
Participants
  Alkaline Phosphatase: number analyzed (Participants) | 8 | 0 | 218 | 61 | 3 | 13 | 39 | 43
  Alkaline Phosphatase: Cohort A - Baseline Value: Low | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase: Cohort B - Baseline Value: Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Alkaline Phosphatase: Cohort A - Baseline Value: Normal | 5 | 0 | 210 | 0 | 0 | 0 | 38 | 0
  Alkaline Phosphatase: Cohort B - Baseline Value: Normal | 0 | 0 | 0 | 61 | 0 | 4 | 0 | 35
  Alkaline Phosphatase: Cohort A - Baseline Value: High | 0 | 0 | 4 | 0 | 3 | 0 | 0 | 0
  Alkaline Phosphatase: Cohort B - Baseline Value: High | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 4
  Alkaline Phosphatase: Cohort A - Baseline Value: Missing | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Alkaline Phosphatase: Cohort B - Baseline Value: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase: number analyzed (Participants) | 0 | 1 | 207 | 67 | 21 | 6 | 40 | 43
  Alanine Aminotransferase: Cohort A - Baseline Value: Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase: Cohort B - Baseline Value: Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase: Cohort A - Baseline Value: Normal | 0 | 0 | 197 | 0 | 7 | 0 | 35 | 0
  Alanine Aminotransferase: Cohort B - Baseline Value: Normal | 0 | 1 | 0 | 67 | 0 | 2 | 0 | 42
  Alanine Aminotransferase: Cohort A - Baseline Value: High | 0 | 0 | 9 | 0 | 14 | 0 | 4 | 0
  Alanine Aminotransferase: Cohort B - Baseline Value: High | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1
  Alanine Aminotransferase: Cohort A - Baseline Value: Missing | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Alanine Aminotransferase: Cohort B - Baseline Value: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase: number analyzed (Participants) | 12 | 0 | 199 | 61 | 12 | 10 | 45 | 46
  Aspartate Aminotransferase: Cohort A - Baseline Value: Low | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase: Cohort B - Baseline Value: Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase: Cohort A - Baseline Value: Normal | 8 | 0 | 193 | 0 | 4 | 0 | 43 | 0
  Aspartate Aminotransferase: Cohort B - Baseline Value: Normal | 0 | 0 | 0 | 60 | 0 | 4 | 0 | 45
  Aspartate Aminotransferase: Cohort A - Baseline Value: High | 0 | 0 | 4 | 0 | 8 | 0 | 1 | 0
  Aspartate Aminotransferase: Cohort B - Baseline Value: High | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 1
  Aspartate Aminotransferase: Cohort A - Baseline Value: Missing | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
  Aspartate Aminotransferase: Cohort B - Baseline Value: Missing | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Bilirubin: number analyzed (Participants) | 1 | 0 | 200 | 70 | 28 | 4 | 39 | 43
  Bilirubin: Cohort A - Baseline Value: Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin: Cohort B - Baseline Value: Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin: Cohort A - Baseline Value: Normal | 1 | 0 | 194 | 0 | 22 | 0 | 33 | 0
  Bilirubin: Cohort B - Baseline Value: Normal | 0 | 0 | 0 | 69 | 0 | 2 | 0 | 41
  Bilirubin: Cohort A - Baseline Value: High | 0 | 0 | 5 | 0 | 6 | 0 | 5 | 0
  Bilirubin: Cohort B - Baseline Value: High | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2
  Bilirubin: Cohort A - Baseline Value: Missing | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Bilirubin: Cohort B - Baseline Value: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium: number analyzed (Participants) | 26 | 1 | 223 | 83 | 1 | 0 | 18 | 33
  Calcium: Cohort A - Baseline Value: Low | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium: Cohort B - Baseline Value: Low | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Calcium: Cohort A - Baseline Value: Normal | 25 | 0 | 219 | 0 | 0 | 0 | 18 | 0
  Calcium: Cohort B - Baseline Value: Normal | 0 | 1 | 0 | 81 | 0 | 0 | 0 | 32
  Calcium: Cohort A - Baseline Value: High | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
  Calcium: Cohort B - Baseline Value: High | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Calcium: Cohort A - Baseline Value: Missing | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Calcium: Cohort B - Baseline Value: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: number analyzed (Participants) | 2 | 5 | 231 | 71 | 19 | 8 | 16 | 33
  Creatinine: Cohort A - Baseline Value: Low | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0
  Creatinine: Cohort B - Baseline Value: Low | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
  Creatinine: Cohort A - Baseline Value: Normal | 1 | 0 | 223 | 0 | 9 | 0 | 15 | 0
  Creatinine: Cohort B - Baseline Value: Normal | 0 | 2 | 0 | 66 | 0 | 2 | 0 | 32
  Creatinine: Cohort A - Baseline Value: High | 0 | 0 | 4 | 0 | 8 | 0 | 0 | 0
  Creatinine: Cohort B - Baseline Value: High | 0 | 0 | 0 | 3 | 0 | 6 | 0 | 1
  Creatinine: Cohort A - Baseline Value: Missing | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
  Creatinine: Cohort B - Baseline Value: Missing | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Glucose: number analyzed (Participants) | 0 | 2 | 178 | 39 | 73 | 43 | 17 | 33
  Glucose: Cohort A - Baseline Value: Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose: Cohort B - Baseline Value: Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose: Cohort A - Baseline Value: Normal | 0 | 0 | 155 | 0 | 19 | 0 | 9 | 0
  Glucose: Cohort B - Baseline Value: Normal | 0 | 2 | 0 | 25 | 0 | 14 | 0 | 16
  Glucose: Cohort A - Baseline Value: High | 0 | 0 | 20 | 0 | 53 | 0 | 7 | 0
  Glucose: Cohort B - Baseline Value: High | 0 | 0 | 0 | 13 | 0 | 29 | 0 | 17
  Glucose: Cohort A - Baseline Value: Missing | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 0
  Glucose: Cohort B - Baseline Value: Missing | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Potassium: number analyzed (Participants) | 5 | 2 | 237 | 78 | 7 | 1 | 19 | 36
  Potassium: Cohort A - Baseline Value: Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium: Cohort B - Baseline Value: Low | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Potassium: Cohort A - Baseline Value: Normal | 5 | 0 | 226 | 0 | 7 | 0 | 18 | 0
  Potassium: Cohort B - Baseline Value: Normal | 0 | 2 | 0 | 75 | 0 | 0 | 0 | 35
  Potassium: Cohort A - Baseline Value: High | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0
  Potassium: Cohort B - Baseline Value: High | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
  Potassium: Cohort A - Baseline Value: Missing | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0
  Potassium: Cohort B - Baseline Value: Missing | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Urea Nitrogen: number analyzed (Participants) | 3 | 0 | 235 | 58 | 15 | 24 | 15 | 35
  Urea Nitrogen: Cohort A - Baseline Value: Low | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Cohort B - Baseline Value: Low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Cohort A - Baseline Value: Normal | 1 | 0 | 222 | 0 | 8 | 0 | 12 | 0
  Urea Nitrogen: Cohort B - Baseline Value: Normal | 0 | 0 | 0 | 54 | 0 | 8 | 0 | 25
  Urea Nitrogen: Cohort A - Baseline Value: High | 0 | 0 | 11 | 0 | 7 | 0 | 2 | 0
  Urea Nitrogen: Cohort B - Baseline Value: High | 0 | 0 | 0 | 4 | 0 | 16 | 0 | 10
  Urea Nitrogen: Cohort A - Baseline Value: Missing | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
  Urea Nitrogen: Cohort B - Baseline Value: Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Changes From Baseline in Electrocardiogram (ECG) Parameters (Safety Outcome Measure)
Time Frame: Changes in ECG pre-drug dosing and within 1-2 hours post-dosing
Population: The Safety Set includes all participants who received any amount of 18F-DCFPyL and have reported data (i.e., some participants had missing ECG measurements).
Measure: Count of Participants; unit: Participants
Groups:
- High Risk Prostate Cancer (Cohort A) - Baseline ECG: High risk prostate cancer participants planned for radical prostatectomy with pelvic lymph node dissection (Cohort A) were enrolled to receive a single dose of 9 mCi (333 MBq) IV injection of 18F-DCFPyL, followed by PET/CT imaging acquired 1-2 hours post-PyL injection. Participants had a 12-lead electrocardiogram (ECG) taken on the day of dosing, prior to dosing.
- High Risk Prostate Cancer (Cohort A) - Post-dosing ECG: High risk prostate cancer participants planned for radical prostatectomy with pelvic lymph node dissection (Cohort A) were enrolled to receive a single dose of 9 mCi (333 MBq) IV injection of 18F-DCFPyL, followed by PET/CT imaging acquired 1-2 hours post-PyL injection. Participants had a 12-lead electrocardiogram (ECG) taken after dosing and prior to imaging.
- Recurrent or Metastatic Prostate Cancer (Cohort B) - Baseline ECG: Participants with presumptive radiologic evidence of prostate cancer recurrence or metastasis on conventional imaging and planned for conventional image-guided biopsy (Cohort B) were enrolled to receive a single dose of 9 mCi (333 MBq) IV injection of 18F-DCFPyL, followed by PET/CT imaging acquired 1-2 hours post-PyL injection.
- Recurrent or Metastatic Prostate Cancer (Cohort B) - Post-dosing ECG: Participants with presumptive radiologic evidence of prostate cancer recurrence or metastasis on conventional imaging and planned for conventional image-guided biopsy (Cohort B) were enrolled to receive a single dose of 9 mCi (333 MBq) IV injection of 18F-DCFPyL, followed by PET/CT imaging acquired 1-2 hours post-PyL injection. Participants had a 12-lead electrocardiogram (ECG) taken after dosing and prior to imaging.
Arm/Group | High Risk Prostate Cancer (Cohort A) - Baseline ECG | High Risk Prostate Cancer (Cohort A) - Post-dosing ECG | Recurrent or Metastatic Prostate Cancer (Cohort B) - Baseline ECG | Recurrent or Metastatic Prostate Cancer (Cohort B) - Post-dosing ECG
Number analyzed (Participants) | 260 | 264 | 114 | 115
Participants
  Normal ECG Evaluation | 159 | 155 | 55 | 51
  Abnormal ECG Evaluation | 101 | 109 | 59 | 64

6. Secondary Outcome: Mean Changes From Baseline in Blood Pressure Post 18F-DCFPyL Dosing (Safety Outcome Measure)
Time Frame: Measured at two intervals on the day of dosing, pre-dosing (baseline) and post-dosing/pre-imaging.
Population: The Safety Set includes all participants who received any amount of 18F-DCFPyL and have reported data (i.e., some participants had missing vital sign measurements).
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- High Risk Prostate Cancer (Cohort A): High risk prostate cancer participants planned for radical prostatectomy with pelvic lymph node dissection (Cohort A) were enrolled to receive a single dose of 9 mCi (333 MBq) IV injection of 18F-DCFPyL, followed by PET/CT imaging acquired 1-2 hours post-PyL injection.
- Recurrent or Metastatic Prostate Cancer (Cohort B): Participants with presumptive radiologic evidence of prostate cancer recurrence or metastasis on conventional imaging and planned for conventional image-guided biopsy (Cohort B) were enrolled to receive a single dose of 9 mCi (333 MBq) IV injection of 18F-DCFPyL, followed by PET/CT imaging acquired 1-2 hours post-PyL injection.
Arm/Group | High Risk Prostate Cancer (Cohort A) | Recurrent or Metastatic Prostate Cancer (Cohort B)
Number analyzed (Participants) | 268 | 117
mm Hg
  Systolic Blood Pressure: Baseline (Actual) | 133.7 (15.99) | 133.6 (19.00)
  Systolic Blood Pressure: Post-dosing (Actual): number analyzed (Participants) | 265 | 114
  Systolic Blood Pressure: Post-dosing (Actual) | 133.7 (16.57) | 132.1 (19.11)
  Systolic Blood Pressure: Change from Baseline: number analyzed (Participants) | 265 | 114
  Systolic Blood Pressure: Change from Baseline | 0.1 (12.30) | -1.3 (11.57)
  Diastolic Blood Pressure: Baseline (Actual) | 79.3 (8.62) | 77.2 (10.16)
  Diastolic Blood Pressure: Post-dosing (Actual): number analyzed (Participants) | 265 | 114
  Diastolic Blood Pressure: Post-dosing (Actual) | 78.5 (9.12) | 76.4 (9.02)
  Diastolic Blood Pressure: Change from Baseline: number analyzed (Participants) | 265 | 114
  Diastolic Blood Pressure: Change from Baseline | -0.7 (7.04) | -0.7 (8.18)

7. Secondary Outcome: Mean Change From Baseline in Heart Rate Post 18F-DCFPyL Dosing (Safety Outcome Measure)
Time Frame: Measured at two intervals on the day of dosing, pre-dosing (baseline) and post-dosing/pre-imaging.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | High Risk Prostate Cancer (Cohort A) | Recurrent or Metastatic Prostate Cancer (Cohort B)
Number analyzed (Participants) | 268 | 117
beats per minute
  Heart Rate: Baseline (Actual) | 70.7 (12.03) | 71.3 (12.94)
  Heart Rate: Post-dosing (Actual): number analyzed (Participants) | 265 | 114
  Heart Rate: Post-dosing (Actual) | 66.4 (10.98) | 67.0 (11.23)
  Heart Rate: Change from Baseline: number analyzed (Participants) | 265 | 114
  Heart Rate: Change from Baseline | -4.4 (6.88) | -4.6 (6.53)

8. Secondary Outcome: Mean Change From Baseline in Respiration Rate Post 18F-DCFPyL Dosing (Safety Outcome Measure)
Time Frame: Measured at two intervals on the day of dosing, pre-dosing (baseline) and post-dosing/pre-imaging.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | High Risk Prostate Cancer (Cohort A) | Recurrent or Metastatic Prostate Cancer (Cohort B)
Number analyzed (Participants) | 265 | 117
breaths per minute
  Respiration Rate: Baseline (Actual) | 16.7 (3.33) | 17.3 (2.16)
  Respiration Rate: Post-dosing (Actual): number analyzed (Participants) | 260 | 114
  Respiration Rate: Post-dosing (Actual) | 16.6 (3.32) | 17.3 (2.28)
  Respiration Rate: Change from Baseline: number analyzed (Participants) | 260 | 114
  Respiration Rate: Change from Baseline | -0.1 (2.03) | 0.0 (2.00)

9. Secondary Outcome: Mean Change From Baseline in Temperature Post 18F-DCFPyL Dosing (Safety Outcome Measure)
Time Frame: Measured at two intervals on the day of dosing, pre-dosing (baseline) and post-dosing/pre-imaging.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | High Risk Prostate Cancer (Cohort A) | Recurrent or Metastatic Prostate Cancer (Cohort B)
Number analyzed (Participants) | 266 | 117
degrees Celsius
  Temperature: Baseline (Actual) | 36.58 (0.433) | 36.56 (0.338)
  Temperature: Post-dosing (Actual): number analyzed (Participants) | 263 | 113
  Temperature: Post-dosing (Actual) | 36.50 (0.479) | 36.59 (0.309)
  Temperature: Change from Baseline: number analyzed (Participants) | 261 | 113
  Temperature: Change from Baseline | -0.08 (0.496) | 0.03 (0.265)

10. Secondary Outcome: Sensitivity of 18F-DCFPyL PET/CT Imaging to Detect Prostate Cancer Within Sites of Metastasis or Local Recurrence Relative to Histopathology in Participants With Recurrent or Metastatic Prostate Cancer (Cohort B)
Description: Sensitivity (True Positive rate) measures the proportion of positives that are correctly identified (i.e., the proportion of those who have some condition (affected) who are correctly identified as having the condition).
Time Frame: Within 28 days of 18F-DCFPyL PET/CT imaging, conventional image-guided biopsy occurred.
Population: Participants with recurrent or metastatic prostate cancer who received 18F-DCFPyL, underwent a conventional image-guided biopsy, and provided an 18F-DCFPyL PET/CT image result and a corresponding histopathology result, along with a conventional image that confirmed the location of the histopathology sample.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Recurrent or Metastatic Prostate Cancer (Cohort B): Participants with presumptive radiologic evidence of prostate cancer recurrence or metastasis on conventional imaging and planned for conventional image-guided biopsy were enrolled to receive a single dose of 9 mCi (333 MBq) IV injection of 18F-DCFPyL, followed by PET/CT imaging acquired 1-2 hours post-PyL injection.
Arm/Group | Recurrent or Metastatic Prostate Cancer (Cohort B)
Number analyzed (Participants) | 93
percentage of participants
  Central Reader 1: number analyzed (Participants) | 92
  Central Reader 1 | 98.6 [91.60 to 100.00]
  Central Reader 2 | 95.8 [87.81 to 99.04]
  Central Reader 3: number analyzed (Participants) | 92
  Central Reader 3 | 92.9 [83.98 to 97.28]

11. Secondary Outcome: Comparison of Detection Rates for Lesion Counts By Location and Overall Between 18F-DCFPyL PET/CT and Conventional Imaging
Description: The number of lesions detected on imaging categorized as bone, visceral/soft tissue, lymph nodes, and the prostate gland will be determined by each of the central imaging core lab independent readers. The sum of lesions per participant per tissue type and overall will be computed for each participant based on each reader's lesion count. This will be calculated from the 18F-DCFPyL PET/CT scan results as well as the conventional imaging results.
Time Frame: Within 1-2 hours of 18F-DCFPyL dosing, a whole body PET/CT scan will be taken
Population: The Evaluable Set consisted of high risk cancer participants (Cohort A) who received 18F-DCFPyL and had a prostatectomy or lymphadenectomy, and participants with recurrent or metastatic prostate cancer (Cohort B) who received 18F-DCFPyL and had a conventional image-guided biopsy, and had an 18F-DCFPyL PET/CT imaging result and a corresponding histology result.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A - Conventional Imaging: High risk prostate cancer participants planned for radical prostatectomy with pelvic lymph node dissection (Cohort A) had baseline CT or MRI images provided to the independent central imaging core lab for assessment by a single reader for prostate cancer detection. The conventional central reader did not assess 18F-DCFPyL PET/CT images. The conventional imaging reader was blinded to local radiology assessments, clinical information, and 18F-DCFPyL PET/CT scans for study participants.
- Cohort A - 18F-DCFPyL PET/CT: Reader 1; Cohort A - 18F-DCFPyL PET/CT: Reader 2; Cohort A - 18F-DCFPyL PET/CT: Reader 3; Cohort B - 18F-DCFPyL PET/CT: Reader 1; Cohort B - 18F-DCFPyL PET/CT: Reader 2; Cohort B - 18F-DCFPyL PET/CT: Reader 3: One of 3 independent core lab readers assigned to assess the 18F-DCFPyL PET/CT image for prostate cancer. The reader was blinded to local radiology assessments, clinical information, conventional imaging scans, and the 18F-DCFPyL PET/CT imaging reads performed by other independent core lab readers.
- Cohort B - Conventional Imaging: Participants with presumptive radiologic evidence of prostate cancer recurrence or metastasis on conventional imaging and planned for conventional image-guided biopsy (Cohort B) had baseline CT or MRI images provided to the independent central imaging core lab for assessment by a single reader for prostate cancer detection. The conventional central reader did not assess 18F-DCFPyL PET/CT images. The conventional imaging reader was blinded to local radiology assessments, clinical information, and 18F-DCFPyL PET/CT scans for study participants.
Arm/Group | Cohort A - Conventional Imaging | Cohort A - 18F-DCFPyL PET/CT: Reader 1 | Cohort A - 18F-DCFPyL PET/CT: Reader 2 | Cohort A - 18F-DCFPyL PET/CT: Reader 3 | Cohort B - Conventional Imaging | Cohort B - 18F-DCFPyL PET/CT: Reader 1 | Cohort B - 18F-DCFPyL PET/CT: Reader 2 | Cohort B - 18F-DCFPyL PET/CT: Reader 3
Number analyzed (Participants) | 252 | 252 | 252 | 252 | 92 | 93 | 93 | 93
Participants
  Tissue Site: Bone: number analyzed (Participants) | 251 | 252 | 252 | 252 | 92 | 93 | 93 | 93
  Tissue Site: Bone: Number of Lesions: 0 | 239 | 234 | 247 | 237 | 37 | 22 | 28 | 23
  Tissue Site: Bone: Number of Lesions: 1-2 | 9 | 17 | 4 | 13 | 20 | 21 | 24 | 22
  Tissue Site: Bone: Number of Lesions: 3-4 | 0 | 1 | 1 | 2 | 8 | 10 | 4 | 10
  Tissue Site: Bone: Number of Lesions: 5-6 | 2 | 0 | 0 | 0 | 1 | 3 | 5 | 2
  Tissue Site: Bone: Number of Lesions: >6 | 1 | 0 | 0 | 0 | 26 | 37 | 32 | 36
  Tissue Site: Visceral/Soft Tissue: number analyzed (Participants) | 251 | 252 | 252 | 252 | 92 | 93 | 93 | 93
  Tissue Site: Visceral/Soft Tissue: Number of Lesions: 0 | 233 | 241 | 249 | 240 | 72 | 71 | 73 | 64
  Tissue Site: Visceral/Soft Tissue: Number of Lesions: 1-2 | 16 | 11 | 3 | 12 | 13 | 15 | 14 | 20
  Tissue Site: Visceral/Soft Tissue: Number of Lesions: 3-4 | 1 | 0 | 0 | 0 | 3 | 2 | 1 | 4
  Tissue Site: Visceral/Soft Tissue: Number of Lesions: 5-6 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0
  Tissue Site: Visceral/Soft Tissue: Number of Lesions: >6 | 1 | 0 | 0 | 0 | 2 | 4 | 3 | 5
  Tissue Site: Lymph Nodes: number analyzed (Participants) | 251 | 252 | 252 | 252 | 92 | 93 | 93 | 93
  Tissue Site: Lymph Nodes: Number of Lesions: 0 | 157 | 216 | 226 | 218 | 37 | 38 | 37 | 38
  Tissue Site: Lymph Nodes: Number of Lesions: 1-2 | 39 | 28 | 19 | 25 | 18 | 11 | 16 | 10
  Tissue Site: Lymph Nodes: Number of Lesions: 3-4 | 10 | 5 | 4 | 5 | 8 | 7 | 13 | 10
  Tissue Site: Lymph Nodes: Number of Lesions: 5-6 | 16 | 3 | 3 | 3 | 7 | 8 | 4 | 8
  Tissue Site: Lymph Nodes: Number of Lesions: >6 | 29 | 0 | 0 | 1 | 22 | 29 | 23 | 27
  Tissue Site: Prostate Gland: number analyzed (Participants) | 250 | 252 | 252 | 252 | 91 | 93 | 93 | 93
  Tissue Site: Prostate Gland: Number of Lesions: 0 | 162 | 5 | 5 | 14 | 79 | 64 | 69 | 63
  Tissue Site: Prostate Gland: Number of Lesions: 1-2 | 88 | 199 | 209 | 204 | 12 | 20 | 22 | 30
  Tissue Site: Prostate Gland: Number of Lesions: 3-4 | 0 | 38 | 33 | 31 | 0 | 6 | 1 | 0
  Tissue Site: Prostate Gland: Number of Lesions: 5-6 | 0 | 10 | 4 | 3 | 0 | 1 | 0 | 0
  Tissue Site: Prostate Gland: Number of Lesions: >6 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
  Tissue Site: All: Number of Lesions: 0 | 109 | 3 | 5 | 14 | 14 | 3 | 11 | 7
  Tissue Site: All: Number of Lesions: 1-2 | 75 | 174 | 196 | 175 | 11 | 15 | 17 | 14
  Tissue Site: All: Number of Lesions: 3-4 | 16 | 55 | 38 | 47 | 8 | 10 | 9 | 8
  Tissue Site: All: Number of Lesions: 5-6 | 17 | 9 | 10 | 11 | 9 | 9 | 10 | 11
  Tissue Site: All: Number of Lesions: >6 | 35 | 11 | 3 | 5 | 50 | 56 | 46 | 53
Statistical Analysis 1: Comparison: Cohort A - Conventional Imaging vs Cohort A - 18F-DCFPyL PET/CT: Reader 1; Tissue Site: Bone; Test type: Superiority; p = 0.1097, Fisher Exact
Statistical Analysis 2: Comparison: Cohort A - Conventional Imaging vs Cohort A - 18F-DCFPyL PET/CT: Reader 2; Tissue Site: Bone; Test type: Superiority; p = 0.1087, Fisher Exact
Statistical Analysis 3: Comparison: Cohort A - Conventional Imaging vs Cohort A - 18F-DCFPyL PET/CT: Reader 3; Tissue Site: Bone; Test type: Superiority; p = 0.1949, Fisher Exact
Statistical Analysis 4: Comparison: Cohort B - Conventional Imaging vs Cohort B - 18F-DCFPyL PET/CT: Reader 1; Tissue Site: Bone; Test type: Superiority; p = 0.1315, Fisher Exact
Statistical Analysis 5: Comparison: Cohort B - Conventional Imaging vs Cohort B - 18F-DCFPyL PET/CT: Reader 2; Tissue Site: Bone; Test type: Superiority; p = 0.1977, Fisher Exact
Statistical Analysis 6: Comparison: Cohort B - Conventional Imaging vs Cohort B - 18F-DCFPyL PET/CT: Reader 3; Tissue Site: Bone; Test type: Superiority; p = 0.2149, Fisher Exact
Statistical Analysis 7: Comparison: Cohort A - Conventional Imaging vs Cohort A - 18F-DCFPyL PET/CT: Reader 1; Tissue Site: Visceral/Soft tissue; Test type: Superiority; p = 0.2582, Fisher Exact
Statistical Analysis 8: Comparison: Cohort A - Conventional Imaging vs Cohort A - 18F-DCFPyL PET/CT: Reader 2; Tissue Site: Visceral/Soft tissue; Test type: Superiority; p = 0.0009, Fisher Exact
Statistical Analysis 9: Comparison: Cohort A - Conventional Imaging vs Cohort A - 18F-DCFPyL PET/CT: Reader 3; Tissue Site: Visceral/Soft tissue; Test type: Superiority; p = 0.3588, Fisher Exact
Statistical Analysis 10: Comparison: Cohort B - Conventional Imaging vs Cohort B - 18F-DCFPyL PET/CT: Reader 1; Tissue Site: Visceral/Soft tissue; Test type: Superiority; p = 0.8791, Fisher Exact
Statistical Analysis 11: Comparison: Cohort B - Conventional Imaging vs Cohort B - 18F-DCFPyL PET/CT: Reader 2; Tissue Site: Visceral/Soft tissue; Test type: Superiority; p = 0.9457, Fisher Exact
Statistical Analysis 12: Comparison: Cohort B - Conventional Imaging vs Cohort B - 18F-DCFPyL PET/CT: Reader 3; Tissue Site: Visceral/Soft tissue; Test type: Superiority; p = 0.2705, Fisher Exact
Statistical Analysis 13: Comparison: Cohort A - Conventional Imaging vs Cohort A - 18F-DCFPyL PET/CT: Reader 1; Tissue Type: Lymph nodes; Test type: Superiority; p < 0.0001, Chi-squared
Statistical Analysis 14: Comparison: Cohort A - Conventional Imaging vs Cohort A - 18F-DCFPyL PET/CT: Reader 2; Tissue Type: Lymph nodes; Test type: Superiority; p < 0.0001, Chi-squared
Statistical Analysis 15: Comparison: Cohort A - Conventional Imaging vs Cohort A - 18F-DCFPyL PET/CT: Reader 3; Tissue Type: Lymph nodes; Test type: Superiority; p < 0.0001, Chi-squared
Statistical Analysis 16: Comparison: Cohort B - Conventional Imaging vs Cohort B - 18F-DCFPyL PET/CT: Reader 1; Tissue Type: Lymph nodes; Test type: Superiority; p = 0.5933, Chi-squared
Statistical Analysis 17: Comparison: Cohort B - Conventional Imaging vs Cohort B - 18F-DCFPyL PET/CT: Reader 2; Tissue Type: Lymph nodes; Test type: Superiority; p = 0.7094, Chi-squared
Statistical Analysis 18: Comparison: Cohort B - Conventional Imaging vs Cohort B - 18F-DCFPyL PET/CT: Reader 3; Tissue Type: Lymph nodes; Test type: Superiority; p = 0.5424, Chi-squared
Statistical Analysis 19: Comparison: Cohort A - Conventional Imaging vs Cohort A - 18F-DCFPyL PET/CT: Reader 1; Tissue Site: Prostate Gland; Test type: Superiority; p < 0.0001, Chi-squared
Statistical Analysis 20: Comparison: Cohort A - Conventional Imaging vs Cohort A - 18F-DCFPyL PET/CT: Reader 2; Tissue Site: Prostate Gland; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 21: Comparison: Cohort A - Conventional Imaging vs Cohort A - 18F-DCFPyL PET/CT: Reader 3; Tissue Site: Prostate Gland; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 22: Comparison: Cohort B - Conventional Imaging vs Cohort B - 18F-DCFPyL PET/CT: Reader 1; Tissue Site: Prostate Gland; Test type: Superiority; p = 0.0038, Fisher Exact
Statistical Analysis 23: Comparison: Cohort B - Conventional Imaging vs Cohort B - 18F-DCFPyL PET/CT: Reader 2; Tissue Site: Prostate Gland; Test type: Superiority; p = 0.0647, Fisher Exact
Statistical Analysis 24: Comparison: Cohort B - Conventional Imaging vs Cohort B - 18F-DCFPyL PET/CT: Reader 3; Tissue Site: Prostate Gland; Test type: Superiority; p = 0.0021, Chi-squared
Statistical Analysis 25: Comparison: Cohort A - Conventional Imaging vs Cohort A - 18F-DCFPyL PET/CT: Reader 1; Tissue Site: All; Test type: Superiority; p < 0.0001, Chi-squared
Statistical Analysis 26: Comparison: Cohort A - Conventional Imaging vs Cohort A - 18F-DCFPyL PET/CT: Reader 2; Tissue Site: All; Test type: Superiority; p < 0.0001, Chi-squared
Statistical Analysis 27: Comparison: Cohort A - Conventional Imaging vs Cohort A - 18F-DCFPyL PET/CT: Reader 3; Tissue Site: All; Test type: Superiority; p < 0.0001, Chi-squared
Statistical Analysis 28: Comparison: Cohort B - Conventional Imaging vs Cohort B - 18F-DCFPyL PET/CT: Reader 1; Tissue Site: All; Test type: Superiority; p = 0.0815, Chi-squared
Statistical Analysis 29: Comparison: Cohort B - Conventional Imaging vs Cohort B - 18F-DCFPyL PET/CT: Reader 2; Tissue Site: All; Test type: Superiority; p = 0.7507, Chi-squared
Statistical Analysis 30: Comparison: Cohort B - Conventional Imaging vs Cohort B - 18F-DCFPyL PET/CT: Reader 3; Tissue Site: All; Test type: Superiority; p = 0.5620, Chi-squared

12. Secondary Outcome: Positive Predictive Value (PPV) of 18F-DCFPyL PET/CT to Predict Prostate Cancer Within the Prostate Gland of High Risk Prostate Cancer Participants (Cohort A)
Description: Positive Predictive Value (PPV) is based on a 18F-DCFPyL PET/CT image result and a histopathology result. The PPV is determined from the number of true positives (positive 18F-DCFPyL image and a positive histopathology result for prostate cancer) divided by the number of participants with a positive 18F-DCFPyL image.
Time Frame: Within 28 days of imaging, radical prostatectomy with pelvic lymph node dissection will occur.
Population: The Evaluable Set of high risk prostate cancer participants (Cohort A) includes those who received 18F-DCFPyL, had a prostatectomy or lymphadenectomy, and had a 18F-DCFPyL PET/CT image result and a corresponding histopathology result.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High Risk Prostate Cancer (Cohort A)
Number analyzed (Participants) | 247
percentage of participants
  Central Reader 1 | 100.0 [98.1 to 100.0]
  Central Reader 2 | 100.0 [98.1 to 100.0]
  Central Reader 3 | 100.0 [98.1 to 100.0]

13. Secondary Outcome: Negative Predictive Value (NPV) of 18F-DCFPyL PET/CT to Predict Prostate Cancer Within the Prostate Gland of High Risk Prostate Cancer Participants (Cohort A)
Description: Negative Predictive Value (NPV) is based on a 18F-DCFPyL PET/CT image result and a histopathology result. The NPV is determined from the number of true negatives (negative 18F-DCFPyL image and a negative histopathology result for prostate cancer) divided by the number of participants with a negative 18F-DCFPyL image.
Time Frame: Within 28 days of imaging, radical prostatectomy with pelvic lymph node dissection will occur.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High Risk Prostate Cancer (Cohort A)
Number analyzed (Participants) | 247
percentage of participants
  Central Reader 1 | 0 [NA to NA] — NPV was 0 - no participant had negative histology in the prostate.
  Central Reader 2 | 0 [NA to NA] — NPV was 0 - no participant had negative histology in the prostate.
  Central Reader 3 | 0 [NA to NA] — NPV was 0 - no participant had negative histology in the prostate.

14. Secondary Outcome: Positive Predictive Value (PPV) of 18F-DCFPyL PET/CT to Predict Prostate Cancer Within the Lymph Nodes of High Risk Prostate Cancer Participants (Cohort A)
Description: as for outcome 12
Time Frame: Within 28 days of imaging, radical prostatectomy with pelvic lymph node dissection will occur.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High Risk Prostate Cancer (Cohort A)
Number analyzed (Participants) | 252
percentage of participants
  Central Reader 1 | 86.7 [69.7 to 95.3]
  Central Reader 2 | 90.5 [69.9 to 98.6]
  Central Reader 3 | 78.1 [63.8 to 92.5]

15. Secondary Outcome: Negative Predictive Value (NPV) of 18F-DCFPyL PET/CT to Predict Prostate Cancer Within the Lymph Nodes of High Risk Prostate Cancer Participants (Cohort A)
Description: as for outcome 13
Time Frame: Within 28 days of imaging, radical prostatectomy with pelvic lymph node dissection will occur.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High Risk Prostate Cancer (Cohort A)
Number analyzed (Participants) | 252
percentage of participants
  Central Reader 1 | 83.8 [78.9 to 88.6]
  Central Reader 2 | 81.4 [76.4 to 86.4]
  Central Reader 3 | 83.2 [78.2 to 88.1]

16. Secondary Outcome: Positive Predictive Value (PPV) of 18F-DCFPyL PET/CT Imaging to Predict Prostate Cancer Within Sites of Local Recurrence and Other Metastatic Lesions in Participants With Recurrent or Metastatic Prostate Cancer (Cohort B)
Description: Positive Predictive Value (PPV) is based on a 18F-DCFPyL PET/CT image result and a histopathology result. The PPV is determined from the number of true positives (positive 18F-DCFPyL image and a positive histopathology result for prostate cancer) divided by the number of participants with a positive 18F-DCFPyL PET/CT image.
Time Frame: Within 28 days of 18F-DCFPyL PET/CT imaging, conventional image-guided biopsy will occur.
Population: The Evaluable Set consisted of participants in Cohort B who received 18F-DCFPyl, had an 18F-DCFPyL PET/CT imaging result, had a conventional image-guided biopsy and a corresponding histology result.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Recurrent or Metastatic Prostate Cancer (Cohort B)
Number analyzed (Participants) | 93
percentage of participants
  Central Reader 1: number analyzed (Participants) | 92
  Central Reader 1 | 81.2 [72.9 to 89.5]
  Central Reader 2 | 81.9 [73.7 to 90.2]
  Central Reader 3: number analyzed (Participants) | 92
  Central Reader 3 | 87.8 [80.4 to 95.3]

17. Secondary Outcome: Peak Plasma Concentration (Cmax) of 18F-DCFPyL in a Subset of Participants
Time Frame: Samples were collected at 0, 5, 15, 30, 60, 120, 240, 360, and 480 minutes after administration of 18F-DCFPyL.
Population: Ten (10) participants from a single investigational site with high risk localized prostate cancer scheduled to undergo radical prostatectomy with pelvic lymph node dissection (Cohort A) agreed and were consented to participate in the PK portion of the study.
Measure: Mean (Standard Deviation); unit: µCi/mL
Groups:
- Pharmacokinetic Subset of High Risk Prostate Cancer Participants (Cohort A): A subset of high risk prostate cancer participants planned for radical prostatectomy with pelvic lymph node dissection (Cohort A) participated in the pharmacokinetic portion of the study.
Arm/Group | Pharmacokinetic Subset of High Risk Prostate Cancer Participants (Cohort A)
Number analyzed (Participants) | 10
µCi/mL | 0.43 (0.088)

18. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of 18F-DCFPyL in a Subset of Participants
Time Frame: Samples were collected at 0, 5, 15, 30, 60, 120, 240, 360, and 480 minutes after administration of 18F-DCFPyL.
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: h*μCi/ml
Arm/Group | Pharmacokinetic Subset of High Risk Prostate Cancer Participants (Cohort A)
Number analyzed (Participants) | 10
h*μCi/ml | 0.82 (0.143)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from Day 1 after 18F-DCFPyL administration through the day prior to prostatectomy, lymphadenectomy or a change in planned protocol procedure (Cohort A); if a participant did not have a procedure, TEAEs were collected for up to 10 days after 18F-DCFPyL administration. For participants in Cohort B, TEAEs were collected from Day 1 after 18F-DCFPyL administration through 28 days after biopsy.
Arm/Group | High Risk Prostate Cancer (Cohort A) | Recurrent or Metastatic Prostate Cancer (Cohort B)
All-Cause Mortality (participants affected / at risk) | 0/268 | 0/117
Serious Adverse Events (participants affected / at risk) | 1/268 | 6/117
Other Adverse Events (participants affected / at risk) | 26/268 | 1/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Risk Prostate Cancer (Cohort A) (N=268) | Recurrent or Metastatic Prostate Cancer (Cohort B) (N=117)
coronary artery disease (Cardiac disorders) | 1 | 1
atrial fibrillation (Cardiac disorders) | 0 | 1
Lower gastrointestinal haemmorhage (Gastrointestinal disorders) | 0 | 1
pyelonephritis, acute (Infections and infestations) | 0 | 1
hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
spinal cord compression (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Risk Prostate Cancer (Cohort A) (N=268) | Recurrent or Metastatic Prostate Cancer (Cohort B) (N=117)
dysgeusia (Nervous system disorders) | 9 | 1
headache (Nervous system disorders) | 9 | 0
fatigue (General disorders) | 5 | 0
diarrhea (Gastrointestinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study results cannot be published before the earlier of a multi-site publication; or 18 months after the end of the Study at all sites; or confirmation by Sponsor that there will be no multi-site publication. The proposed publication must be submitted to Sponsor at least 60 days prior to publication so that Sponsor can delete Sponsor Confidential Information (other than Study results) and obtain a further 60 days to file on any invention disclosed in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT02981368/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/68/NCT02981368/SAP_001.pdf